CLINICAL TRIAL: NCT07005791
Title: 基于人工智能的视神经鞘超声视频构建肺癌软脑膜转移患者颅内压预测模型及多模态临床预后模型的双中心临床研究
Brief Title: AI-Based Ultrasound Prediction Model for Intracranial Pressure and Prognosis in Lung Cancer Patients With Leptomeningeal Metastasis: A Dual-Center Study
Status: Not yet recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Nanjing University (Other); Nanjing Jiangning Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-LCYJ-PY-60
Record Dates: First submitted 2024-10-21; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2024-09

CONDITIONS: Lung Cancer (NSCLC); Leptomeningeal Metastasis; Intracranial Pressure
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Meningeal Carcinomatosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study focuses on developing an innovative, artificial intelligence-based model using optic nerve sheath ultrasound videos to predict intracranial pressure in lung cancer patients with leptomeningeal metastasis. The study also aims to create a multimodal clinical prognosis model that can help improve patient outcomes. By analyzing ultrasound data from patients at two major medical centres, the research seeks to provide more accurate and early predictions of complications related to elevated intracranial pressure, ultimately improving treatment and management strategies for these patients.

ELIGIBILITY:
Inclusion Criteria:

1- Age: Participants must be aged 18 years or older. 2、Diagnosis: Patients must have a histologically confirmed diagnosis of non-small cell lung cancer (NSCLC) with clinically or pathologically confirmed leptomeningeal metastases (LM), and at least one measurable lesion.

3、Lumbar Puncture and Intrathecal Chemotherapy: Patients must have undergone lumbar puncture and intrathecal chemotherapy in the study center.

4、ECOG Performance Status: Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 3.

5、Blood Tests: Neutrophil count ≥ 1.5 × 10⁹/L. Hemoglobin ≥ 9 g/dL. Platelet count ≥ 100 × 10⁹/L. 6、Biochemical Tests: Total bilirubin ≤ 1.5 times the upper limit of normal (ULN). AST (aspartate aminotransferase) and ALT (alanine aminotransferase) < 1.5 times ULN.

Creatinine clearance ≥ 60 ml/min. 7、No Significant Bleeding or Thrombosis: Patients must not have significant bleeding symptoms, bleeding disorders, or active thrombosis.

8、Reproductive Health: Women of childbearing age must use appropriate contraception and have a negative pregnancy test prior to enrollment.

9、Informed Consent: All patients must have signed the informed consent form and be willing to comply with the study procedures and follow-up schedule.

Exclusion Criteria:

* 1、Histological Type: Patients with squamous cell carcinoma or small cell lung cancer are excluded.

  2、Recent Radiotherapy: Patients who have received local radiotherapy for intracranial lesions within the past two weeks are excluded.

  3、ECOG Performance Status: Patients with an ECOG performance score greater than 3 are excluded.

  4、Uncontrolled Seizures: Patients with uncontrolled seizures are excluded. 5、Other Tumor History: Patients with a current or past history of other tumors are excluded.

  6、Bleeding or Thrombotic Disorders: Patients with known hereditary or acquired bleeding or thrombotic tendencies (e.g., hemophilia, coagulation disorders, thrombocytopenia) or with abnormal coagulation function (INR > 2.0, PT > 16s) are excluded. Those on thrombolytic or anticoagulant therapy are also excluded, except for patients on preventive doses of low-dose aspirin or low-molecular-weight heparin.

  7、Recent Trauma or Surgery: Patients with a history of severe trauma or surgery within the last month, or significant bleeding events within the past three months, are excluded.

  8、Severe Organ Dysfunction: Patients with severe hepatic or renal dysfunction, HIV infection, HCV infection, asthma, or uncontrolled cerebrovascular disease are excluded.

  9、Pregnancy and Breastfeeding: Pregnant or breastfeeding women are excluded. Women of childbearing age must test negative for pregnancy within seven days prior to enrollment.

  10、Thrombotic Events: Patients with arterial or venous thrombotic events (e.g., stroke, transient ischemic attack, brain hemorrhage, deep vein thrombosis, or pulmonary embolism) within the past six months are excluded.

  11、Safety Concerns: Any other conditions or factors that the investigator deems unsuitable for inclusion, including issues that might compromise the patient's safety or compliance, will result in exclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Primary Diagnosis: Patients diagnosed with non-small cell lung cancer (NSCLC), confirmed through histopathological examination.
  2. Leptomeningeal Metastases (LM): Patients with clinically or pathologically confirmed LM, a serious complication of NSCLC characterized by cancer spread to the membranes surrounding the brain and spinal cord.
  3. Age Range: Patients aged 18 years or older.
  4. ECOG Performance Status: Patients must have an ECOG score of 3 or lower, indicating varying degrees of functionality but generally not bedridden.
  5. Intrathecal Chemotherapy: The study focuses on patients undergoing lumbar puncture and intrathecal chemotherapy as part of their treatment.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the Intracranial Pressure (ICP) Prediction Model and Efficacy of the Prognostic Model | Half an hour before the lumbar puncture
  Accuracy of the Intracranial Pressure (ICP) Prediction Model: This involves constructing a prediction model for ICP based on optic nerve sheath diameter (ONSD) and other ultrasound measurements (e.g., optic disk height, ODH). The model's accuracy will be evaluated by comparing the predicted ICP values with those obtained through lumbar puncture, using metrics such as the area under the ROC curve (AUC), sensitivity, and specificity.
  Efficacy of the Prognostic Model: This model will predict clinical outcomes such as progression-free survival (PFS) and overall survival (OS) based on multimodal data, including clinical and imaging data. The predictive performance will be assessed using the C-index and other statistical measures to determine its effectiveness in forecasting patient outcomes.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Jiangning Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing Drum-tower Hospital Affiliated to Medical College of Nanjing University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No